CLINICAL TRIAL: NCT00656799
Title: A Single Center, Open-Label Trial in Subjects With Severe Renal Impairment Evaluating the Dialysability of the Sugammadex-Rocuronium Complex
Brief Title: Dialysis of Sugammadex in Participants With Severe Renal Impairment (Study 19.4.333) (P05773)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05773; 2007-006934-33 (EudraCT Number)
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Results first posted 2013-07-31 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-02

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Sugammadex; Rocuronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sugammadex (Experimental): IV single bolus dose of 4.0 mg/kg sugammadex
  Interventions: Drug: sugammadex; Drug: Rocuronium

INTERVENTIONS:
Drug: sugammadex — At 15 minutes after administration of rocuronium, an IV single bolus dose of 4.0 mg/kg sugammadex was administered.
  Other Names: Org 25969; SCH 900616; MK-8616; Bridion®
Drug: Rocuronium — After achieving stable anesthesia an IV single bolus dose of 0.6 mg/kg rocuronium was administered
  Other Names: Rocuronium bromide; Esmeron®

SUMMARY:
The clinical trial objectives were to evaluate the dialysability of the sugammadex-rocuronium complex; it's safety and efficacy in participants with severe renal impairment.

DETAILED DESCRIPTION:
The current trial was designed to evaluate the dialysability of the sugammadex-rocuronium complex in participants with severe renal impairment. A dose of 4.0 mg/kg sugammadex was administered 15 minutes after administration of 0.6 mg/kg rocuronium. Blood and dialysate samples were collected before, during and after hemodialysis/filtration, for calculation of clearance of sugammadex-rocuronium complex and assessment of rebound.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* American Society of Anesthesiologists (ASA) Class >=4
* Creatinine clearance (CLCR) < 30 mL/min and clinical indication for dialysis
* Hospitalization at Intensive Care Unit (ICU) and scheduled for a (surgical) procedure under general anesthesia requiring neuromuscular relaxation with the use of rocuronium
* Scheduled for a (surgical) procedure in supine position
* Written informed consent (of the legal representative)

Exclusion Criteria:

* Known or suspected to have neuromuscular disorders impairing neuromuscular blockade and/or significant hepatic dysfunction
* Known or suspected to have a (family) history of malignant hyperthermia
* Known or suspected to have an allergy to narcotics, muscle relaxants or other medication used during general anesthesia
* Have already participated in a sugammadex trial
* Have participated in another clinical trial, not preapproved by NV Organon, within 30 days of study entry
* Females who are pregnant*
* Females who are breast-feeding * In females pregnancy will be excluded both from medical history and by a human chorionic gonadotropin (hCG) test within 24 hours before surgery except in females who are not of childbearing potential, i.e. at least 2 years menopausal or have undergone tubal ligation or an hysterectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

REFERENCES:
- [Result] Cammu G, Van Vlem B, van den Heuvel M, Stet L, el Galta R, Eloot S, Demeyer I. Dialysability of sugammadex and its complex with rocuronium in intensive care patients with severe renal impairment. Br J Anaesth. 2012 Sep;109(3):382-90. doi: 10.1093/bja/aes207. Epub 2012 Jun 24. PMID 22732111

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugammadex: Intravenous (IV) single bolus dose of 4.0 mg/kg sugammadex
Period: Overall Study
Arm/Group | Sugammadex
Started | 6
Completed | 4
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Sugammadex
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 76 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Clearance of Sugammadex by Dialysis as Measured by the Reduction Ratio (RR)
Description: Starting on Day 1 dialysis was performed on four separate occasions using a Fresenius 40008H hemodialyzer, with a hemodiafilter standard helixone membrane FX 600. Dialysate samples were collected before, and after hemodialysis, with concentrations of sugammadex determined using a liquid chromatographic assay with mass spectrometric detection. The clearance of sugammadex at each dialysis session was calculated by measuring the ratio of plasma concentration at the end of dialysis, average duration of 6 hours, compared with that immediately before the start of dialysis, called the RR.
Time Frame: Up to day 7
Population: All subjects pharmacokinetically evaluable consisting of all participants who received a dose of sugammadex and had at least one efficacy measurement
Measure: Mean (Standard Deviation); unit: Reduction Ratio
Arm/Group | Sugammadex
Number analyzed (Participants) | 6
Reduction Ratio
  First Dialysis (n=5) | 0.687 (0.113)
  Second Dialysis (n=6) | 0.566 (0.150)
  Third Dialysis (n=4) | 0.516 (0.232)
  Fourth Dialysis (n=4) | 0.532 (0.144)

2. Secondary Outcome: Number of Participants With Pre-treatment Adverse Events (AEs)
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body, whether or not related to the use of a product.
Time Frame: Screening up to Day 1
Population: All Subjects Treated (AST) consisting of participants who received a dose of sugammadex
Measure: Number; unit: participants
Arm/Group | Sugammadex
Number analyzed (Participants) | 6
participants | 1

3. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A SAE is any untoward medical occurrence that at any dose results in the following: death, is life threatening, requires in-patient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, or is a congenital anomaly/birth defect
Time Frame: Up to day 7
Population: AST consisting of all participants who received a dose of sugammadex
Measure: Number; unit: participants
Arm/Group | Sugammadex
Number analyzed (Participants) | 6
participants | 2

4. Secondary Outcome: Number of Participants With Medical Device (Near) Incidents
Description: A medical device (near) incident is defined as an occurrence due to inaccurate or inadequate labeling/instructions, or information supplied with a medical device; or malfunction, deterioration or recall of a medical device that could lead to death or serious deterioration in health.
Time Frame: Up to day 7
Population: AST consisting of all participants who received a dose of sugammadex
Measure: Number; unit: participants
Arm/Group | Sugammadex
Number analyzed (Participants) | 6
participants | 0

5. Secondary Outcome: Vital Sign: Mean Systolic Blood Pressure
Description: Systolic blood pressure was measured at the following time points: screening, before rocuronium treatment, before sugammadex treatment, at 2, 5, 10, 20 minutes post-sugammadex treatment, and the day after surgery
Time Frame: Screening up to 1 day after surgery
Population: AST consisting of all participants who received a dose of sugammadex
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Sugammadex
Number analyzed (Participants) | 6
mm Hg
  Screening | 124.2 (19.2)
  Pre-Rocuronium | 106.3 (25.2)
  Baseline pre-sugammadex | 105.5 (20.4)
  2 minutes post-sugammadex | 105.0 (11.5)
  5 minutes post-sugammadex | 103.2 (10.0)
  10 minutes post-sugammadex | 98.0 (10.9)
  30 minutes post-sugammadx | 92.8 (21.3)
  Post-anesthetic | 146.3 (26.7)

6. Secondary Outcome: Vital Sign: Mean Diastolic Blood Pressure
Description: Diastolic blood pressure was measured at the following time points: screening, before rocuronium treatment, before sugammadex treatment, at 2, 5, 10, 20 minutes post-sugammadex treatment, and the day after surgery
Time Frame: Screening up to 1 day after surgery
Population: AST consisting of all participants who received a dose of sugammadex
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Sugammadex
Number analyzed (Participants) | 6
mm Hg
  Screening | 58.2 (6.2)
  Pre-Rocuronium | 51.2 (13.6)
  Baseline pre-sugammadex | 45.2 (13.3)
  2 minutes post-sugammadex | 46.5 (12.3)
  5 minutes post-sugammadex | 44.5 (12.1)
  10 minutes post-sugammadex | 46.8 (8.9)
  30 minutes post-sugammadex | 43.7 (9.4)
  Post-anesthetic | 67.8 (13.2)

7. Secondary Outcome: Vital Sign: Mean Heart Rate
Description: Heart rate was measured at the following time points: screening, before rocuronium treatment, before sugammadex treatment, at 2, 5, 10, 20 minutes post-sugammadex treatment, and the day after surgery
Time Frame: Screening up to 1 day after surgery
Population: AST consisting of all participants who received a dose of sugammadex
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Sugammadex
Number analyzed (Participants) | 6
Beats per minute
  Screening | 81.7 (22.6)
  Pre-Rocuronium | 78.0 (21.4)
  Baseline pre-sugammadex | 83.7 (21.4)
  2 minutes post-sugammadex | 81.0 (20.8)
  5 minutes post-sugammadex | 80.5 (20.4)
  10 minutes post-sugammadex | 80.2 (20.4)
  30 minutes post-sugammadex | 77.8 (20.1)
  Post-anesthetic | 71.8 (11.1)

8. Secondary Outcome: Number of Participants With Physical Examinations
Description: Physical examinations were to be conducted at screening, on Day 1 and 7 days after surgery
Time Frame: Screening up to day 7
Population: AST consisting of all participants who received a dose of sugammadex
Measure: Number; unit: participants
Arm/Group | Sugammadex
Number analyzed (Participants) | 6
participants
  Screening | 6
  Peri-procedural (Day 1) | 6
  Day 7 | 0

9. Secondary Outcome: Number of Participants With Reoccurrence of Neuromuscular Blockade at Day 1
Description: Neuromuscular function was monitored by applying repetitive train of four (TOF) electrical stimulations to the ulnar nerve every 15 seconds and assessing the magnitudes (heights) of the first twitch (T1) and fourth twitch (T4) response at the adductor pollicis muscle with a TOF-Watch® SX. Stimulation continued until the T4/T1 ratio reached at least 0.9. Higher T4/T1 ratios represent greater recovery from neuromuscular blockade; with a value of 1.0 representing full recovery. Reoccurrence of neuromuscular blockade is defined as a decline in the T4/T1 ratio from >= 0.9 to < 0.8 in at least three consecutive measurements.
Time Frame: Day 1
Population: AST consisting of all screened participants who received a dose of sugammadex
Measure: Number; unit: participants
Arm/Group | Sugammadex
Number analyzed (Participants) | 6
participants | 0

10. Secondary Outcome: Number of Participants With Events Due to Possible Interaction of Sugammadex With Endo-/Exogenous Compounds Other Than Rocuronium
Description: Evidence of AEs due to possible interaction of sugammadex with endogenous compounds or with exogenous compounds other than rocuronium
Time Frame: Day 1
Population: AST consisting of all participants who received a dose of sugammadex
Measure: Number; unit: participants
Arm/Group | Sugammadex
Number analyzed (Participants) | 6
participants | 0

11. Secondary Outcome: Number of Participants With Pregnancies at 30 Days Post-dose
Description: Pregnancies reported by means of a Pregnancy Reporting Form, consist of pregnant female participants or pregnant female partners of male participants
Time Frame: Up to 30 days post -dose
Population: AST consisting of all participants who received a dose of sugammadex
Measure: Number; unit: participants
Arm/Group | Sugammadex
Number analyzed (Participants) | 6
participants | 0

12. Secondary Outcome: Time From Start of Administration of Sugammadex to Recovery of T4/T1 Ratio to 0.9
Description: Neuromuscular function was monitored by applying repetitive train of four (TOF) electrical stimulations to the ulnar nerve every 15 seconds and assessing the magnitudes (heights) of the first twitch (T1) and fourth twitch (T4) response at the adductor pollicis muscle with a TOF-Watch® SX. Stimulation continued until the T4/T1 ratio reached at least 0.9. Higher T4/T1 ratios represent greater recovery from neuromuscular blockade; with a value of 1.0 representing full recovery.
Time Frame: Day 1
Population: Intent To Treat (ITT) group consisting of participants who received a dose of sugammadex and had at least one efficacy measurement
Measure: Geometric Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Sugammadex
Number analyzed (Participants) | 6
Minutes | 5.11 [3.06 to 8.53]

13. Secondary Outcome: Time From Start of Administration of Sugammadex to Recovery of T4/T1 Ratio to 0.8
Description: Neuromuscular function was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds and assessing the magnitudes (heights) of the T1 and T4 response at the adductor pollicis muscle with a TOF-Watch® SX. Stimulation continued until the T4/T1 ratio reached at least 0.8. Higher T4/T1 ratios represent greater recovery from neuromuscular blockade; with a value of 1.0 representing full recovery.
Time Frame: Day 1
Population: ITT group consisting of participants who received a dose of sugammadex and had at least one efficacy measurement
Measure: Geometric Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Sugammadex
Number analyzed (Participants) | 6
Minutes | 4.05 [2.36 to 6.93]

14. Secondary Outcome: Time From Start of Administration of Sugammadex to Recovery of T4/T1 Ratio to 0.7
Description: Neuromuscular function was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds and assessing the magnitudes (heights) of the T1 and T4 response at the adductor pollicis muscle with a TOF-Watch® SX. Stimulation continued until the T4/T1 ratio reached at least 0.7. Higher T4/T1 ratios represent greater recovery from neuromuscular blockade; with a value of 1.0 representing full recovery.
Time Frame: Day 1
Population: ITT group consisting of participants who received a dose of sugammadex and had at least one efficacy measurement
Measure: Geometric Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Sugammadex
Number analyzed (Participants) | 6
Minutes | 3.41 [1.90 to 6.15]

15. Primary Outcome: Clearance of Rocuronium by Dialysis as Measured by the Reduction Ratio (RR)
Description: Starting on Day 1 dialysis was performed on four separate occasions using a Fresenius 40008H hemodialyzer, with a hemodiafilter standard helixone membrane FX 600. Dialysate samples were collected before, and after hemodialysis, with concentrations of rocuronium determined using a liquid chromatographic assay with mass spectrometric detection. The clearance of rocuronium at each dialysis session was calculated by measuring the ratio of plasma concentration at the end of dialysis, average duration of 6 hours, compared with that immediately before the start of dialysis, called the RR.
Time Frame: Up to Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Reduction Ratio
Arm/Group | Sugammadex
Number analyzed (Participants) | 6
Reduction Ratio
  First Dialysis (n=5) | 0.750 (0.0786)
  Second Dialysis (n=6) | 0.625 (0.144)
  Third Dialysis (n=4) | 0.521 (0.0489)
  Fourth Dialysis (n=4) | 0.458 (0.115)

16. Primary Outcome: Rate of Clearance of Sugammadex From Blood
Description: Starting on Day 1 dialysis was performed on four separate occasions using a Fresenius 40008H hemodialyzer, with a hemodiafilter standard helixone membrane FX 600. Blood samples were collected from ports in the arterial and venous tubing of the dialyzer before, during and after an average of 6 hours of hemodialysis. The concentrations of sugammadex were determined using a liquid chromatographic assay with mass spectrometric detection. The clearance rate from blood at each dialysis session was assessed by averaging across all available collection time points.
Time Frame: Up to day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Sugammadex
Number analyzed (Participants) | 6
mL/min
  First Dialysis (n=5) | 79.1 (19.0)
  Second Dialysis (n=6) | 76.5 (19.6)
  Third Dialysis (n=4) | 72.4 (18.4)
  Fourth Dialysis (n=4) | 83.4 (16.5)

17. Primary Outcome: Rate of Clearance of Rocuronium From Blood
Description: Starting on Day 1 dialysis was performed on four separate occasions using a Fresenius 40008H hemodialyzer, with a hemodiafilter standard helixone membrane FX 600. Blood samples were collected from ports in the arterial and venous tubing of the dialyzer before, during and after an average of 6 hours of hemodialysis. The concentrations of rocuronium were determined using a liquid chromatographic assay with mass spectrometric detection. The clearance rate from blood at each dialysis session was assessed by averaging across all available collection time points.
Time Frame: Up to Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Sugammadex
Number analyzed (Participants) | 6
mL/min
  First Dialysis (n=5) | 80.2 (15.2)
  Second Dialysis (n=6) | 86.3 (14.1)
  Third Dialysis (n=4) | 94.1 (14.8)
  Fourth Dialysis (n=3) | 94.8 (9.68)

18. Primary Outcome: Rate of Clearance of Sugammadex From Dialysate
Description: Starting on Day 1 dialysis was performed on four separate occasions using a Fresenius 40008H hemodialyzer, with a hemodiafilter standard helixone membrane FX 600. Dialysate samples were collected from a port in the outflow of the dialyzer before, during and after an average of 6 hours of hemodialysis. The concentrations of sugammadex were determined using a liquid chromatographic assay with mass spectrometric detection. The clearance rate from dialysate at each dialysis session was assessed by averaging across all available collection time points.The data from the fourth dialysis are not presented as they were not calculable.
Time Frame: Up to day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Sugammadex
Number analyzed (Participants) | 6
mL/min
  First Dialysis (n=5) | 63.0 (8.74)
  Second Dialysis (n=6) | 65.1 (7.06)
  Third Dialysis (n=4) | 66.8 (13.2)

19. Primary Outcome: Rate of Clearance of Rocuronium From Dialysate
Description: Starting on Day 1 dialysis was performed on four separate occasions using a Fresenius 40008H hemodialyzer, with a hemodiafilter standard helixone membrane FX 600. Dialysate samples were collected from a port in the outflow of the dialyzer before, during and after an average of 6 hours of hemodialysis. The concentrations of rocuronium were determined using a liquid chromatographic assay with mass spectrometric detection. The clearance rate from dialysate at each dialysis session was assessed by averaging across all available collection time points.
Time Frame: Up to Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Sugammadex
Number analyzed (Participants) | 6
mL/min
  First Dialysis (n=5) | 75.1 (5.81)
  Second Dialysis (n=6) | 97.2 (32.4)
  Third Dialysis (n=4) | 110 (36.4)
  Fourth Dialysis (n=4) | 95.3 (19.2)

ADVERSE EVENTS:
Time Frame: Up to 7 days after administration of sugammadex
Arm/Group | Sugammadex
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex (N=6)
Cardiac failure (Cardiac disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex (N=6)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Decubitis ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In case a proposed publication contains reference to an invention owned by the sponsor or to which the sponsor otherwise has rights, the sponsor may request a reasonable suspension of the publication.